CLINICAL TRIAL: NCT00332163
Title: A Phase 2, Open-label, Randomized Clinical Trial of Skin Toxicity Treatment in Subjects Receiving Second-line FOLFIRI or Irinotecan Only Chemotherapy Concomitantly With Panitumumab
Brief Title: Skin Toxicity Treatment in Metastatic Colorectal Cancer (mCRC) Patients Receiving Panitumumab + Irinotecan-based Therapy
Acronym: STEPP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20050184
Record Dates: First submitted 2006-05-31; First posted 2006-06-01 (Estimated); Results first posted 2016-02-23 (Estimated); Last update posted 2016-02-23 (Estimated); Status verified 2016-01

CONDITIONS: Metastatic Colorectal Cancer; Skin Rash; Skin Toxicities; Colon Cancer; Colorectal Cancer
Keywords: STEPP; STEP; STEEP; mCRC; Skin Toxicities; Skin Rash; Metastatic Colorectal Cancer; Anti-EGFr Skin Rash; colon cancer; colorectal cancer; rectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Exanthema; Colonic Neoplasms; Rectal Neoplasms | interventions — Panitumumab; Irinotecan; IFL protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pre-emptive Skin Treatment (Experimental): Participants received either FOLFIRI and panitumumab 6 mg/kg once every 2 weeks (Q2W) or irinotecan and panitumumab 9 mg/kg once every 3 weeks (Q3W), and pre-emptive skin treatment which included skin moisturizer, sunscreen, 1% hydrocortisone cream, and an oral antibiotic for 6 weeks starting 24 hours prior to chemotherapy.
  Interventions: Biological: Panitumumab; Drug: Irinotecan; Drug: FOLFIRI; Drug: Pre-emptive Skin Treatment
- Reactive Skin Treatment (Experimental): Participants received either FOLFIRI and panitumumab 6 mg/kg Q2W or irinotecan and panitumumab 9 mg/kg Q3W. Participants were treated for each individual skin toxicity occurrence according to prespecified guidelines and based on the type and severity. Treatment could include emollient, sunscreen, topical or oral steroids, antibiotics, or antihistamines, as required.
  Interventions: Biological: Panitumumab; Drug: Irinotecan; Drug: FOLFIRI; Drug: Reactive Skin Treatment

INTERVENTIONS:
Biological: Panitumumab — Administered by intravenous infusion
  Other Names: Vectibix
Drug: Irinotecan — Recommended dosage regimen and administration of irinotecan was based on local standard of care, the package insert, and institutional guidelines.
Drug: FOLFIRI — Chemotherapy consisting of irinotecan with infusional 5-fluorouracil and leucovorin. Recommended dosage regimen and administration of FOLFIRI was based on local standard of care, the package insert for each product, and institutional guidelines.
Drug: Pre-emptive Skin Treatment — Pre-emptive skin treatment included a skin moisturizer (eg, Lubriderm), sunscreen (free of paraaminobenzoic acid (PABA), skin protection factor (SPF) 15 or higher, ultraviolet-A (UV-A), and UV-B protection), topical steroid (1% hydrocortisone cream) and oral antibiotic (doxycycline, 100 mg twice daily).
  Arms: Pre-emptive Skin Treatment
Drug: Reactive Skin Treatment — Treatment was based on symptoms and severity and may have included an emollient (eg, Lubriderm, Vaseline), sunscreen (SPF ≥ 15), oral antibiotic (eg, doxycycline, ciprofloxacin, cefadroxil, amoxicillin/clavulanic acid), topical steroid (hydrocortisone cream), topical antibiotic (clindamycin), oral systemic steroid, topical medical treatment (eg, silver sulfadiazine, Silvadene), topical antihistamine or oral antihistamine (hydroxyzine)
  Arms: Reactive Skin Treatment

SUMMARY:
A comparison of prophylactic treatment with reactive treatment for skin toxicity observed in patients with metastatic colorectal cancer (mCRC) who are receiving second-line irinotecan-based chemotherapy concomitantly with panitumumab.

ELIGIBILITY:
Inclusion Criteria:

* Patients with unresectable metastatic adenocarcinoma of the colon or rectum that cannot, in the opinion of the investigator, be cured by surgical resection at the time of randomization;
* Patients who have failed first line treatment containing fluoropyrimidine and oxaliplatin based chemotherapy with or without bevacizumab for mCRC.

Exclusion Criteria:

• Prior irinotecan use for the treatment of mCRC.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2006-04; Primary Completion 2008-01 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Background] Lacouture ME, Mitchell EP, Piperdi B, Pillai MV, Shearer H, Iannotti N, Xu F, Yassine M. Skin toxicity evaluation protocol with panitumumab (STEPP), a phase II, open-label, randomized trial evaluating the impact of a pre-Emptive Skin treatment regimen on skin toxicities and quality of life in patients with metastatic colorectal cancer. J Clin Oncol. 2010 Mar 10;28(8):1351-7. doi: 10.1200/JCO.2008.21.7828. Epub 2010 Feb 8. PMID 20142600
- [Derived] Weeraratne D, Chen A, Pennucci JJ, Wu CY, Zhang K, Wright J, Perez-Ruixo JJ, Yang BB, Kaliyaperumal A, Gupta S, Swanson SJ, Chirmule N, Starcevic M. Immunogenicity of panitumumab in combination chemotherapy clinical trials. BMC Clin Pharmacol. 2011 Nov 9;11:17. doi: 10.1186/1472-6904-11-17. PMID 22070868
- [Derived] Mitchell EP, Piperdi B, Lacouture ME, Shearer H, Iannotti N, Pillai MV, Xu F, Yassine M. The efficacy and safety of panitumumab administered concomitantly with FOLFIRI or Irinotecan in second-line therapy for metastatic colorectal cancer: the secondary analysis from STEPP (Skin Toxicity Evaluation Protocol With Panitumumab) by KRAS status. Clin Colorectal Cancer. 2011 Dec;10(4):333-9. doi: 10.1016/j.clcc.2011.06.004. Epub 2011 Oct 14. PMID 22000810
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants enrolled at 36 sites in the United States between 17 April 2006 and 28 September 2007.
Pre-assignment Details: Participants were stratified to receive either a FOLFIRI and panitumumab regimen or an irinotecan and panitumumab regimen based on the investigator's discretion according to local standard of care. Participants were then randomized to receive either a pre-emptive skin treatment or reactive skin treatment regimen for a 6-week skin treatment period.
Period: Overall Study
Arm/Group | Pre-emptive Skin Treatment | Reactive Skin Treatment
Started | 48 | 47
Received Treatment | 48 | 47
Completed | 48 | 47
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pre-emptive Skin Treatment | Reactive Skin Treatment | Total
Number analyzed (Participants) | 48 | 47 | 95
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.6 (12.7) | 61.1 (9.9) | 60.8 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 21 | 37
  Male | 32 | 26 | 58
Race/Ethnicity, Customized [Number; unit: participants]
  White or Caucasian | 34 | 40 | 74
  Black or African American | 6 | 5 | 11
  Hispanic or Latino | 5 | 1 | 6
  Asian | 2 | 0 | 2
  Native Hawaiian or other Pacific Islander | 1 | 0 | 1
  Other | 0 | 1 | 1
Chemotherapy Stratification [Number; unit: participants]
  FOLFIRI + Panitumumab Q2W | 28 | 27 | 55
  Irinotecan + Panitumumab Q3W | 20 | 20 | 40

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Specific Grade 2 or Higher Skin Toxicities During the 6-week Skin Treatment Period
Description: Skin toxicities were assessed by the study clinician and graded according to the modified Common Toxicity Criteria for Adverse Events (CTCAE) v.3.0 Dermatology Toxicity Grading criteria, on a scale from Grade 1 (mild) to 4 (life-threatening). The specific skin toxicities of interest were pruritus, acneiform dermatitis, skin desquamation (also described as skin exfoliation), exfoliative dermatitis, paronychia, nail disorder, skin fissures, skin laceration, pruritic rash, pustular rash, skin infection, skin ulceration, and local infection.
Time Frame: 6 weeks
Population: Primary analysis set (all randomized participants who provided informed consent before protocol-specific procedures and who received at least 1 dose of panitumumab)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pre-emptive Skin Treatment | Reactive Skin Treatment
Number analyzed (Participants) | 48 | 47
percentage of participants | 29 [16 to 42] | 62 [48 to 76]
Statistical Analysis 1: Comparison: Pre-emptive Skin Treatment vs Reactive Skin Treatment; Test type: Superiority or Other; Difference = -33, 95% CI 2-sided [-51 to -14] — Difference = Pre-emptive - Reactive

2. Secondary Outcome: Percentage of Participants With Any Grade 2 or Higher Skin Toxicity of Any Type During the 6-week Skin Treatment Period
Description: The percentage of participants who developed at least 1 incidence of ≥ grade 2 skin toxicities of any type during the 6-week skin treatment period. Analysis of this endpoint was based on adverse event data associated with the "Skin and Subcutaneous Tissue Disorders" system organ class. Adverse events were graded according to the National Cancer Institute (NCI) CTCAE version 3.0.
Time Frame: 6 weeks
Population: Primary Analysis Set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pre-emptive Skin Treatment | Reactive Skin Treatment
Number analyzed (Participants) | 48 | 47
percentage of participants | 40 [26 to 53] | 62 [48 to 76]
Statistical Analysis 1: Comparison: Pre-emptive Skin Treatment vs Reactive Skin Treatment; Test type: Superiority or Other; Difference = -22, 95% CI 2-sided [-42 to -3] — Difference = Pre-emptive - Reactive

3. Secondary Outcome: Time to First Occurrence of Specific Grade 2 or Higher Skin Toxicities of Interest
Description: The time to the first occurrence of specific grade 2 or higher skin toxicities of interest was defined as the time from the first dose of panitumumab to the date of first occurrence of specific ≥ grade 2 skin toxicities of interest. Participants who did not experience specific skin-related toxicities were censored at their last skin toxicity assessment during the skin toxicity assessment period. Skin toxicities were assessed by the study clinician and graded according to the modified CTCAE v.3.0 Dermatology Toxicity Grading criteria, on a scale from Grade 1 (mild) to 4 (life-threatening). The specific skin toxicities of interest were pruritus, acneiform dermatitis, skin desquamation (also described as skin exfoliation), exfoliative dermatitis, paronychia, nail disorder, skin fissures, skin laceration, pruritic rash, pustular rash, skin infection, skin ulceration, and local infection.
Time Frame: 6 weeks
Population: Primary Analysis Set
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Pre-emptive Skin Treatment | Reactive Skin Treatment
Number analyzed (Participants) | 48 | 47
weeks | NA [NA to NA] — Not reached due to the low number of events | 2.1 [2.1 to 6.3]
Statistical Analysis 1: Comparison: Pre-emptive Skin Treatment vs Reactive Skin Treatment; Test type: Superiority or Other; Hazard Ratio (HR) = 0.4, 95% CI 2-sided [0.2 to 0.7] — Hazard ratio estimated from a Cox Proportional Hazards regression model with an indicator for treatment (pre-emptive vs. reactive), stratified by chemotherapy stratum (Q2W vs Q3W)

4. Secondary Outcome: Most Severe Specific Grade 2 or Higher Skin Toxicities of Interest
Description: The percentage of participants with a most severe grade of 2, 3 or 4 specific skin toxicity of interest reported during the 6-week skin treatment period. Skin toxicities were assessed by the study clinician and graded according to the modified CTCAE v.3.0 Dermatology Toxicity Grading criteria, on a scale from Grade 1 (mild) to 4 (life-threatening). The specific skin toxicities of interest were pruritus, acneiform dermatitis, skin desquamation (also described as skin exfoliation), exfoliative dermatitis, paronychia, nail disorder, skin fissures, skin laceration, pruritic rash, pustular rash, skin infection, skin ulceration, and local infection.
Time Frame: 6 weeks
Population: Primary Analysis Set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pre-emptive Skin Treatment | Reactive Skin Treatment
Number analyzed (Participants) | 48 | 47
percentage of participants
  Grade 2 | 23 [11 to 35] | 40 [26 to 54]
  Grade 3 | 6 [0 to 13] | 21 [10 to 33]
  Grade 4 | 0 [NA to NA] — Could not be estimated as there were no events in this category | 0 [NA to NA] — Could not be estimated as there were no events in this category

5. Secondary Outcome: Time to First Most Severe Specific Grade 2 or Higher Skin Toxicities of Interest
Description: Time to the first most severe grade ≥ 2 of all the specific skin-related toxicities of interest was defined as the time from the first dose of panitumumab to the date of the first occurrence of the most severe specific ≥ grade 2 skin toxicity of interest during the 6-week skin treatment period. Participants who did not experience any specific skin-related toxicity of grade ≥ 2 were censored at their last skin toxicity assessment during the 6-week skin toxicity assessment period. Skin toxicities were assessed by the study clinician and graded according to the modified CTCAE v.3.0 Dermatology Toxicity Grading criteria, on a scale from Grade 1 (mild) to 4 (life-threatening). The specific skin toxicities of interest were pruritus, acneiform dermatitis, skin desquamation (also described as skin exfoliation), exfoliative dermatitis, paronychia, nail disorder, skin fissures, skin laceration, pruritic rash, pustular rash, skin infection, skin ulceration, and local infection.
Time Frame: 6 weeks
Population: Primary Analysis Set
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Pre-emptive Skin Treatment | Reactive Skin Treatment
Number analyzed (Participants) | 48 | 47
weeks | NA [NA to NA] — Could not be estimated due to the low number of events | 2.7 [2.1 to 6.3]
Statistical Analysis 1: Comparison: Pre-emptive Skin Treatment vs Reactive Skin Treatment; Test type: Superiority or Other; Hazard Ratio (HR) = 0.4, 95% CI 2-sided [0.2 to 0.7] — Hazard ratio estimated from a Cox Proportional Hazards regression model with an indicator for treatment (Pre-emptive vs. Reactive) stratified by chemotherapy stratum (Q2W vs Q3W)

6. Secondary Outcome: Percentage of Participants With Panitumumab Dose Reductions Due to the Specific Skin Toxicities of Interest
Time Frame: 6 weeks
Population: Primary Analysis Set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pre-emptive Skin Treatment | Reactive Skin Treatment
Number analyzed (Participants) | 48 | 47
percentage of participants | 6 [0 to 13] | 11 [2 to 19]
Statistical Analysis 1: Comparison: Pre-emptive Skin Treatment vs Reactive Skin Treatment; Test type: Superiority or Other; Difference = -4, 95% CI 2-sided [-16 to 7] — Difference = Pre-emptive - Reactive

7. Secondary Outcome: Response Rate at First Scheduled Assessment
Description: Tumor response was assessed by computed tomography (CT) scan or magnetic resonance imaging (MRI) of the abdomen, pelvis, and all other sites of disease. Disease assessments were performed by central review according to the modified response evaluation criteria in solid tumors (RECIST). Response rate is defined as the percentage of participants with a complete response (CR) or partial response (PR) at the Week 9/10 assessment visit and a corresponding CR or PR confirmed at the Week 13/14 assessment visit for the Q2W/Q3W regimens. CR: Disappearance of all target and non-target lesions and no new lesions. PR: Either the disappearance of all target lesions with persistence of one or more non-target lesion(s) not qualifying for either CR or progressive disease (PD; ≥ 25% increase in lesion size) and no new lesions, or, at least a 30% decrease in the size of target lesions with no progression of existing non-target lesions, and no new lesions.
Time Frame: Week 9 with confirmed response at Week 13 for the FOLFIRI and panitumumab Q2W regimen or at Week 10 with confirmed response at Week 14 for the irinotecan and panitumumab Q3W regimen.
Population: Primary Analysis Set; participants who discontinued prematurely without a post-baseline tumor assessment or with an observed CR or PR at Week 9 or 10 that was not confirmed at Week 13/14 were considered non-responders.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pre-emptive Skin Treatment | Reactive Skin Treatment
Number analyzed (Participants) | 48 | 47
percentage of participants | 6 [0 to 13] | 6 [0 to 13]
Statistical Analysis 1: Comparison: Pre-emptive Skin Treatment vs Reactive Skin Treatment; Test type: Superiority or Other; Difference = 0, 95% CI 2-sided [-10 to 10] — Difference = Pre-emptive - Reactive

8. Secondary Outcome: Best Overall Response Rate
Description: Best overall response rate is defined as the percentage of participants with a complete response (CR) or partial response (PR) while on study. Tumor response was assessed by CT scan or MRI of the abdomen, pelvis, and all other sites of disease. Disease assessments were performed by central review according to the modified RECIST criteria. CR: Disappearance of all target and non-target lesions and no new lesions. PR: Either the disappearance of all target lesions with persistence of one or more non-target lesion(s) not qualifying for either CR or PD (≥ 25% increase in lesion size) and no new lesions, or, at least a 30% decrease in the size of target lesions with no progression of existing non-target lesions, and no new lesions.
Time Frame: Response was assessed at Weeks 9 and 13 and then every 8 weeks for the Q2W regimen, or at Weeks 10, 14, 22 and then every 9 weeks for the Q3W regimen until the end of treatment; median treatment duration was 13 and 17 weeks in each group respectively.
Population: Primary Analysis Set; participants who prematurely discontinued without a post-baseline tumor assessment or with an observed CR or PR that was not confirmed were considered non-responders.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pre-emptive Skin Treatment | Reactive Skin Treatment
Number analyzed (Participants) | 48 | 47
percentage of participants | 15 [5 to 25] | 11 [2 to 19]
Statistical Analysis 1: Comparison: Pre-emptive Skin Treatment vs Reactive Skin Treatment; Test type: Superiority or Other; Difference = 4, 95% CI 2-sided [-9 to 17] — Rate difference = Pre-emptive - Reactive

9. Secondary Outcome: Rate of Disease Control at First Scheduled Assessment
Description: Tumor response was assessed by CT scan or MRI of the abdomen, pelvis, and all other sites of disease. Disease assessments were performed by central review according to the modified response evaluation criteria in solid tumors (RECIST). Disease control rate is defined as the percentage of participants with a CR, PR or stable disease (SD) at the Week 9/10 assessment visit and a corresponding response (CR or PR) confirmed at the Week 13/14 assessment visit for the Q2W/Q3W regimens. SD: Neither sufficient shrinkage or increase in target lesions to qualify for PR or PD, with no progression of non-target lesions and no new lesions.
Time Frame: as for outcome 7
Population: Primary Analysis Set; participants who prematurely discontinued without a postbaseline tumor assessment or with an observed CR or PR at Week 9 or 10 that was not confirmed at Week 13 or 14 were considered non-responders.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pre-emptive Skin Treatment | Reactive Skin Treatment
Number analyzed (Participants) | 48 | 47
percentage of participants | 63 [49 to 76] | 64 [50 to 78]
Statistical Analysis 1: Comparison: Pre-emptive Skin Treatment vs Reactive Skin Treatment; Test type: Superiority or Other; Difference = -1, 95% CI 2-sided [-21 to 18] — Rate difference = Pre-emptive - Reactive

10. Secondary Outcome: Time to Treatment Failure
Description: Time-to-treatment failure is defined as the time from the date of randomization to the first date of any of the following events: discontinuation of study therapy due to any reason (except for complete response and curative surgery), progression of disease, or death due to any cause. Participants who did not discontinue, who were still alive, and who did not have disease progression were censored at the date of last contact. Time to treatment failure was analyzed using the Kaplan-Meier method.
Time Frame: From randomization until the end of study; median time on study was 31 weeks and 41 weeks in each treatment group respectively with a maximum time on study of 97 weeks.
Population: Primary Analysis Set
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pre-emptive Skin Treatment | Reactive Skin Treatment
Number analyzed (Participants) | 48 | 47
months | 3.1 [2.3 to 4.8] | 4.2 [3.2 to 5.3]
Statistical Analysis 1: Comparison: Pre-emptive Skin Treatment vs Reactive Skin Treatment; Test type: Superiority or Other; Hazard Ratio (HR) = 1.3, 95% CI 2-sided [0.9 to 2.0] — [estimate comment as in outcome 5, analysis 1]

11. Secondary Outcome: Time to Progression
Description: Time from the date of randomization to the date of observed disease progression or death due to disease progression. Participants who did not have documented disease progression were censored at the date of last tumor assessment; participants who died for reasons other than disease progression while on study were censored at the date of death. PD: At least a 20% increase in the size of target lesions, recorded since the treatment started, or at least a 25% increase in size of non-target lesions and the lesion(s) measure > 10 mm in one dimension, or the appearance of one or more new lesions.
  Time to progression was analyzed using the Kaplan-Meier method. This analysis excludes any data collected during follow-up for participants who began third-line treatment.
Time Frame: as for outcome 10
Population: Primary Analysis Set
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pre-emptive Skin Treatment | Reactive Skin Treatment
Number analyzed (Participants) | 48 | 47
months | 4.9 [3.1 to 6.4] | 4.1 [2.9 to 6.2]
Statistical Analysis 1: Comparison: Pre-emptive Skin Treatment vs Reactive Skin Treatment; Test type: Superiority or Other; Hazard Ratio (HR) = 0.9, 95% CI 2-sided [0.6 to 1.5] — [estimate comment as in outcome 5, analysis 1]

12. Secondary Outcome: Overall Survival
Description: Overall Survival is defined as the time from the date of randomization to the date of death. Participants who did not die while on study or who were lost-to-follow-up were censored at their last contact date. Overall survival was analyzed using all data regardless of whether it was collected during second- or third-line treatment.
Time Frame: as for outcome 10
Population: Primary Analysis Set
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pre-emptive Skin Treatment | Reactive Skin Treatment
Number analyzed (Participants) | 48 | 47
months | 11.2 [8.3 to 16.1] | 13.6 [9.9 to 19.0]
Statistical Analysis 1: Comparison: Pre-emptive Skin Treatment vs Reactive Skin Treatment; Test type: Superiority or Other; Hazard Ratio (HR) = 1.2, 95% CI 2-sided [0.7 to 2.1] — [estimate comment as in outcome 5, analysis 1]

13. Secondary Outcome: Progression-free Survival
Description: Defined as the time from the date of randomization to the first date of observed disease progression or death due to any cause (whichever comes first). Participants who were alive and had not progressed while on study were censored at the date of last progression-free tumor assessment.
Time Frame: as for outcome 10
Population: Primary Analysis Set
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pre-emptive Skin Treatment | Reactive Skin Treatment
Number analyzed (Participants) | 48 | 47
months | 4.7 [2.9 to 6.0] | 4.1 [2.9 to 6.2]
Statistical Analysis 1: Comparison: Pre-emptive Skin Treatment vs Reactive Skin Treatment; Test type: Superiority or Other; Hazard Ratio (HR) = 1.0, 95% CI 2-sided [0.6 to 1.6] — Hazard ratio is estimated from a Cox Proportional Hazards regression model with an indicator for treatment (Pre-emptive vs. Reactive) stratified by chemotherapy stratum (Q2W vs Q3W)

14. Secondary Outcome: Change From Baseline in Overall Dermatologic Quality of Life Index (DLQI) Score
Description: Skin-related quality of life was assessed using the DLQI. The DLQI questionnaire asks participants to evaluate the degree that their skin condition has affected their quality of life in the last week. Participants answer 10 questions on a scale from 0 (not at all) to 3 (very much); The DLQI score is calculated by summing the scores for all questions, resulting in a maximum of 30 and a minimum of 0; higher scores indicate a more impaired quality of life.
Time Frame: Baseline and Weeks 2, 3, 4, 5, 6 and 7
Population: Patient Reported Outcomes (PRO) Analysis Set (randomized participants who signed informed consent before protocol-specified procedures, received at least 1 dose of panitumumab, with a non-missing baseline overall DLQI score and who had at least 1 post-baseline non-missing overall DLQI score) with available data at each time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pre-emptive Skin Treatment | Reactive Skin Treatment
Number analyzed (Participants) | 46 | 44
units on a scale
  Baseline (n=46, 44) | 0.3 (0.7) | 0.1 (0.3)
  Change from Baseline to Week 2 (n=42, 41) | 0.7 (1.4) | 1.6 (3.7)
  Change from Baseline to Week 3 (n=44, 42) | 1.3 (2.6) | 4.2 (5.8)
  Change from Baseline to Week 4 (n=42, 42) | 1.7 (2.4) | 3.8 (5.4)
  Change from Baseline to Week 5 (n=44, 42) | 1.3 (2.3) | 2.7 (4.2)
  Change from Baseline to Week 6 (n=42, 38) | 1.6 (2.8) | 2.3 (3.9)
  Change from Baseline to Week 7 (n=40, 40) | 2.0 (2.8) | 2.6 (4.4)

ADVERSE EVENTS:
Time Frame: The reporting time frame is from first dose date to 30 days since the last dose date. The median time frames for pre-emptive skin treatment and reactive skin treatment are 3.5 months and 4.7 months, respectively.
Description: Other Adverse Events summarizes the non-serious occurrences of adverse events that exceed the indicated frequency threshold.
Arm/Group | Pre-emptive Skin Treatment | Reactive Skin Treatment
Serious Adverse Events (participants affected / at risk) | 13/48 | 23/47
Other Adverse Events (participants affected / at risk) | 47/48 | 47/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pre-emptive Skin Treatment (N=48) | Reactive Skin Treatment (N=47)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 0 | 3
LEUKOPENIA (Blood and lymphatic system disorders) | 0 | 1
NEUTROPENIA (Blood and lymphatic system disorders) | 0 | 3
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 0 | 1
ATRIAL FIBRILLATION (Cardiac disorders) | 0 | 1
BRADYCARDIA (Cardiac disorders) | 0 | 1
CARDIO-RESPIRATORY ARREST (Cardiac disorders) | 1 | 0
ABDOMINAL PAIN (Gastrointestinal disorders) | 2 | 3
DIARRHOEA (Gastrointestinal disorders) | 2 | 8
GASTROINTESTINAL PERFORATION (Gastrointestinal disorders) | 1 | 0
ILEUS (Gastrointestinal disorders) | 0 | 1
NAUSEA (Gastrointestinal disorders) | 2 | 2
PROCTALGIA (Gastrointestinal disorders) | 1 | 0
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 0 | 1
VOMITING (Gastrointestinal disorders) | 3 | 4
ASTHENIA (General disorders) | 1 | 2
DEATH (General disorders) | 1 | 0
FATIGUE (General disorders) | 1 | 0
NON-CARDIAC CHEST PAIN (General disorders) | 0 | 1
PYREXIA (General disorders) | 1 | 0
CENTRAL LINE INFECTION (Infections and infestations) | 0 | 1
CLOSTRIDIAL INFECTION (Infections and infestations) | 0 | 1
FUNGAL INFECTION (Infections and infestations) | 0 | 1
GASTROENTERITIS (Infections and infestations) | 0 | 1
LOCALISED INFECTION (Infections and infestations) | 0 | 1
SEPSIS (Infections and infestations) | 0 | 2
SEPTIC SHOCK (Infections and infestations) | 0 | 1
STAPHYLOCOCCAL ABSCESS (Infections and infestations) | 1 | 0
STREPTOCOCCAL ABSCESS (Infections and infestations) | 1 | 0
URINARY TRACT INFECTION (Infections and infestations) | 0 | 1
FALL (Injury, poisoning and procedural complications) | 0 | 1
JOINT INJURY (Injury, poisoning and procedural complications) | 0 | 1
WEIGHT DECREASED (Investigations) | 1 | 0
DEHYDRATION (Metabolism and nutrition disorders) | 3 | 9
ELECTROLYTE IMBALANCE (Metabolism and nutrition disorders) | 0 | 1
FAILURE TO THRIVE (Metabolism and nutrition disorders) | 0 | 1
HYPERKALAEMIA (Metabolism and nutrition disorders) | 0 | 1
HYPOKALAEMIA (Metabolism and nutrition disorders) | 0 | 3
HYPOMAGNESAEMIA (Metabolism and nutrition disorders) | 0 | 1
HYPONATRAEMIA (Metabolism and nutrition disorders) | 1 | 0
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 0 | 1
COLON CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
COLON CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
COLORECTAL CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
HEMIPLEGIA (Nervous system disorders) | 0 | 1
SYNCOPE (Nervous system disorders) | 0 | 1
DEPRESSION (Psychiatric disorders) | 0 | 1
MENTAL STATUS CHANGES (Psychiatric disorders) | 1 | 0
RENAL FAILURE (Renal and urinary disorders) | 0 | 1
RENAL FAILURE ACUTE (Renal and urinary disorders) | 0 | 2
URETERIC OBSTRUCTION (Renal and urinary disorders) | 0 | 1
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 | 1
LUNG INFILTRATION (Respiratory, thoracic and mediastinal disorders) | 1 | 0
RASH (Skin and subcutaneous tissue disorders) | 0 | 1
HYPERTENSION (Vascular disorders) | 0 | 1
VENA CAVA THROMBOSIS (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pre-emptive Skin Treatment (N=48) | Reactive Skin Treatment (N=47)
ANAEMIA (Blood and lymphatic system disorders) | 11 | 16
NEUTROPENIA (Blood and lymphatic system disorders) | 9 | 19
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 1 | 6
CONJUNCTIVITIS (Eye disorders) | 3 | 4
EYE IRRITATION (Eye disorders) | 1 | 3
ABDOMINAL PAIN (Gastrointestinal disorders) | 13 | 12
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 3 | 7
CONSTIPATION (Gastrointestinal disorders) | 13 | 14
DIARRHOEA (Gastrointestinal disorders) | 26 | 38
DRY MOUTH (Gastrointestinal disorders) | 3 | 4
DYSPEPSIA (Gastrointestinal disorders) | 6 | 3
FLATULENCE (Gastrointestinal disorders) | 3 | 3
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 1 | 3
NAUSEA (Gastrointestinal disorders) | 32 | 24
PROCTALGIA (Gastrointestinal disorders) | 0 | 3
STOMATITIS (Gastrointestinal disorders) | 11 | 14
VOMITING (Gastrointestinal disorders) | 21 | 16
ASTHENIA (General disorders) | 7 | 7
CHILLS (General disorders) | 5 | 3
FATIGUE (General disorders) | 28 | 27
MUCOSAL INFLAMMATION (General disorders) | 11 | 11
OEDEMA PERIPHERAL (General disorders) | 1 | 6
PAIN (General disorders) | 5 | 1
PYREXIA (General disorders) | 6 | 3
HYPERBILIRUBINAEMIA (Hepatobiliary disorders) | 0 | 3
PARONYCHIA (Infections and infestations) | 8 | 17
RASH PUSTULAR (Infections and infestations) | 13 | 19
SKIN INFECTION (Infections and infestations) | 2 | 5
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 2 | 7
URINARY TRACT INFECTION (Infections and infestations) | 3 | 5
SKIN LACERATION (Injury, poisoning and procedural complications) | 2 | 6
WEIGHT DECREASED (Investigations) | 11 | 12
WHITE BLOOD CELL COUNT DECREASED (Investigations) | 4 | 1
ANOREXIA (Metabolism and nutrition disorders) | 14 | 11
DECREASED APPETITE (Metabolism and nutrition disorders) | 1 | 7
DEHYDRATION (Metabolism and nutrition disorders) | 5 | 13
HYPERKALAEMIA (Metabolism and nutrition disorders) | 0 | 3
HYPOCALCAEMIA (Metabolism and nutrition disorders) | 3 | 5
HYPOKALAEMIA (Metabolism and nutrition disorders) | 9 | 13
HYPOMAGNESAEMIA (Metabolism and nutrition disorders) | 7 | 12
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 1 | 5
BACK PAIN (Musculoskeletal and connective tissue disorders) | 2 | 6
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 1 | 4
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 2 | 6
DIZZINESS (Nervous system disorders) | 5 | 5
HEADACHE (Nervous system disorders) | 1 | 4
NEUROPATHY (Nervous system disorders) | 1 | 4
NEUROPATHY PERIPHERAL (Nervous system disorders) | 6 | 7
ANXIETY (Psychiatric disorders) | 2 | 7
DEPRESSION (Psychiatric disorders) | 3 | 7
INSOMNIA (Psychiatric disorders) | 6 | 10
DYSURIA (Renal and urinary disorders) | 3 | 0
COUGH (Respiratory, thoracic and mediastinal disorders) | 5 | 9
DYSPHONIA (Respiratory, thoracic and mediastinal disorders) | 3 | 1
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 7 | 3
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 3 | 5
PHARYNGOLARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 2 | 4
ALOPECIA (Skin and subcutaneous tissue disorders) | 15 | 13
DERMATITIS ACNEIFORM (Skin and subcutaneous tissue disorders) | 37 | 40
DERMATITIS EXFOLIATIVE (Skin and subcutaneous tissue disorders) | 11 | 12
DRY SKIN (Skin and subcutaneous tissue disorders) | 12 | 9
ERYTHEMA (Skin and subcutaneous tissue disorders) | 9 | 9
NAIL DISORDER (Skin and subcutaneous tissue disorders) | 7 | 10
PRURITUS (Skin and subcutaneous tissue disorders) | 30 | 32
RASH (Skin and subcutaneous tissue disorders) | 3 | 6
RASH ERYTHEMATOUS (Skin and subcutaneous tissue disorders) | 3 | 2
RASH PRURITIC (Skin and subcutaneous tissue disorders) | 19 | 20
SKIN EXFOLIATION (Skin and subcutaneous tissue disorders) | 16 | 19
SKIN FISSURES (Skin and subcutaneous tissue disorders) | 13 | 16
SKIN ULCER (Skin and subcutaneous tissue disorders) | 5 | 4
HYPOTENSION (Vascular disorders) | 2 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.